CLINICAL TRIAL: NCT07305402
Title: A French Multicenter Retrospective Study of Native and Prosthetic Vascular Infections Caused by Coxiella Burnetii (COXIVAS)
Brief Title: Vascular Infections Caused by Coxiella Burnetii
Acronym: COXIVAS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2025/024
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Vascular Infection Caused by C. Burnetii
Keywords: vascular infection; vascular graft infection; vascular endograft infection; Coxiella burnetii

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prosthetic vascular infection due to C. burnetii: Adults with native or prosthetic vascular infection due to C. burnetii

SUMMARY:
high morbidity and mortality. In France, Coxiella burnetii-related vascular infections appear to be increasing, though data remain limited. Two-year mortality reaches 15-18%, mainly due to serious complications such as arterio-digestive fistulas. Diagnosis is often delayed, prognostic factors are poorly defined, and the value of advanced imaging techniques remains insufficiently studied.

DETAILED DESCRIPTION:
Q fever is a worldwide zoonosis that may cause chronic vascular infections with significant morbidity and mortality. In France, the incidence of Coxiella burnetii-related vascular infections appears to be increasing, although published data remain scarce. Reported two-year mortality reaches 15-18%, largely due to severe complications such as arterio-digestive fistulas. Classical risk factors include aortic aneurysm and vascular grafts, but many patients present without clear zoonotic exposure, leading to frequent underdiagnosis. Prognostic factors are poorly defined, apart from the lack of surgical management, which worsens outcomes. Diagnosis is often delayed, and the value of advanced imaging modalities such as 18F-FDG PET/CT or labeled leukocyte scintigraphy remains insufficiently studied.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18yrs old) with native or prosthetic vascular infection due to C. burnetii (Jan 2000 - Dec 2023)
* diagnosis based on CNR vascular Q fever criteria,
* supplemented by MAGIC (Management of Aortic Graft Infection Collaboration) criteria for prosthetic/ - endovascular infections or aortitis/arteritis criteria,
* no objection to reuse of patient data.

Exclusion Criteria:

* patient under legal protection,
* insufficient French language comprehension

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults (≥ 18yrs old) with native or prosthetic vascular infection due to C. burnetii
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
two-year mortality rate | 2 years
  from the time of initial management

SECONDARY OUTCOMES:
Early mortality rate | Day 30
  Early mortality rate (Day 30)
Infection-attributed mortality rate | 2 years
  Infection-attributed mortality rate
Two-year morbidity rate | 2 years
  Two-year morbidity rate
Rate of initial complications | 2 years
  Rate of initial complications
Rate of postoperative complications | 2 years
  Rate of postoperative complications
Diagnostic performance of the different imaging modalities | 2 years
  Diagnostic performance of the different imaging modalities

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No